CLINICAL TRIAL: NCT02996383
Title: Fixation Versus Arthroplasty for Undisplaced Intracapsular Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peterborough and Stamford Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Martyn J Parker, consultant orthopaedic surgeon, Peterborough and Stamford Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R&D/2016/05
Record Dates: First submitted 2016-06-10; First posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Hip Fractures; Undisplaced Intracapsular Hip Fracture
Keywords: arthroplasty
MeSH Terms: conditions — Hip Fractures | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cemented hemiarthroplasty (Active Comparator): Treatment of the fracture by a replacement arthroplasty with a cemented CPT hemiarthroplasty (manafactured by Zimmer company, Warsaw IN, USA) inserted via an anteriolateral approach to the hip
  Interventions: Device: Cemented Hemiarthroplasty
- Internal fixation (Active Comparator): Internal fixation of the fracture with a screw and plate device (Targon FN plate, Aesculap cooperation, Tuttingham, Germany)
  Interventions: Device: Internal fixation

INTERVENTIONS:
Device: Internal fixation — Internal fixation of the fracture with a Targon FN implant (BBraun Ltd, Germany)
  Arms: Internal fixation
Device: Cemented Hemiarthroplasty — Replacement of the femoral head with a cemented hemiarthroplasty
  Arms: Cemented hemiarthroplasty

SUMMARY:
In England each year over 70,000 people fracture their hip. Most of these patients are elderly females with the fracture occurring after a simple trip or stumble. Approximately half of these fractures are classified from their relationship to the hip joint capsule as intracapsular. These fractures are subdivided into those that are displaced and those that are undisplaced. The majority of displaced fractures are treated with a replacement arthroplasty. Current treatment for the undisplaced fractures is generally by internal fixation of the fracture using screws and a plate, although some centres prefer replacement arthroplasty.

A recent randomised study on patients from Norway with undisplaced intracapsular fractures treated with either internal fixation or arthroplasty has just reported reduced complications and re-operations for those patients treated with an arthroplasty. In addition functional results were marginally better for those patients treated with an arthroplasty. Current practice in the UK is generally to treat these fractures by internal fixation. This study aims to see if replacement arthroplasty can indeed lead to the advantages suggested from the Norwegian study.

Patients who satisfy the inclusion criteria and are willing to participate will be randomised to receive either reduction and internal fixation of the fracture with a screw and plate device or alternatively replacement of their femoral head with an artificial hip replacement (hemiarthroplasty). After surgery patients will receive the same treatment as normal and be discharge home when able, with follow-up review in the hip fracture clinic. Subsequent follow-up for the research project is by phone calls from a research nurse who is blinded to the type of treatment that the patient has received. There will be no additional investigations or out-patient follow-up visits for these patients in comparison to normal treatment protocols. Results of the study will ultimately be published in a medical journal.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to Peterborough and Stamford Hospitals NHS Foundation Trust with an undisplaced intracapsular fracture will be considered for inclusion within the study. Patients who lack Capacity for example dementia who are unable to provide informed consent will be included if the assent of their next of kin or legal guardian can be obtained.

Exclusion Criteria:

* • patients who decline to participate or in whom consent or assent is not available

  * patients admitted when MJP is not available to supervise treatment
  * patients with pathological fractures from Paget's disease of bone secondary's from tumour
  * patients with delayed presentation who would be treated conservatively
  * patients considered unfit for either surgical procedure
  * younger patients, aged less than 80 years who are independently mobile and very active will be excluded at treated by internal fixation (the risk of fracture healing complication for this group is less, whilst there is an increased risk of long term complications after arthroplasty

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
regain of mobility using the Parker and Palmer mobility scale | one year
  Assessment is using the Parker and Palmer mobility score (Parker MJ, Palmer CR. A new mobility score for predicting mortality after hip fracture. J Bone Joint Surg Br. 1993;75:797-8.)

CONTACTS AND LOCATIONS:
Locations (1):
- Peterborough and Stamford Hospital NHS Foundation Trust, Peterborough, Cambs, United Kingdom